CLINICAL TRIAL: NCT02406313
Title: Evaluation of the Efficiency of a Therapeutic Education Program in Standardized Thermal Cure for Fibromyalgia Patients
Brief Title: Fibromyalgia Therapeutic Education in Thermal Cure
Acronym: FiETT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00464-43
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTS + ETP (Experimental): Patients following a standardized thermal cure (CTS) follow an additional program called Fibr'eaux (ETP) that consists in discussion groups and physical activities allowing patients to learn how to manage their illness.
  Interventions: Other: CTS; Other: ETP
- CTS alone (Active Comparator): Patients follow a standardized thermal cure that is a sedative, relaxing, antalgic and mobilizing treatment based on muds application, hydrotherapy and physiotherapy. The cure is made of 72 treatments selected among a list including muds application, massages, reeducation in thermal pool, baths and showers.
  Interventions: Other: CTS

INTERVENTIONS:
Other: CTS — Standardized Thermal Cure
Other: ETP — Patient Therapeutic Education
  Arms: CTS + ETP

SUMMARY:
The study evaluates the efficiency, in terms of quality of life improvement, of a patient's therapeutic education program (ETP), based on long term commitment in adapted physical activities carried out during a standardized thermal cure (CTS) for fibromyalgia among patients continuing regular drug treatment or not

DETAILED DESCRIPTION:
Fibromyalgia is a poorly known and understood disease. Patients suffer from pain, fatigue, sleep disorders, anxiety, depression, preventing them from moving and going out, resulting in an alteration of social life. Multiple drugs treatment is frequently used but is burdensome and poorly effective. However, thermal cure proved efficacious to improve quality of life during the cure and beyond. This study aims at demonstrating the added value of a patient's therapeutic education program provided during a thermal cure, a moment where patients are available and receptive to guidance.

ELIGIBILITY:
Inclusion Criteria

* Diagnostic of fibromyalgia done at least 6 months before thermal cure
* Diagnostic of fibromyalgia confirmed by FIRST questionnaire (score 5) during the initial thermal checkup
* Age between 18 and 65 years
* Access to an Internet connection during remote follow-up
* Affiliation to a social security system (recipient or assignee)
* Signed written inform consent form

Exclusion Criteria

* Infectious diseases with ongoing treatment (except for winter upper respiratory tract pathologies)
* Active tumorous pathology
* Concomitant inflammatory rheumatism
* Stage III chronic venous insufficiency with history of phlebitis and/or pulmonary embolism
* Incapacity to receive treatment in hot water ( ≥36°)
* Total incapacity to practice physical activities of therapeutic education program
* Ongoing pregnancy
* Involvement in a structured educational program specific to fibromyalgia during the previous year
* Incapacity to understand French language making the follow up impossible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Month 06 after cure completion
  Change from baseline in quality of life assessed through the self-administered Fibromyalgia Impact Questionnaire (FIQ) month 06 after cure completion.

SECONDARY OUTCOMES:
Change in quality of life | Week 03, Month 03, Month 12
  Average change from baseline in pain intensity measured on a Visual Analogical Scale (VAS)
Responder rate | Week 03, Month 03, Month 06, Month 12
  Rate of patients responding to intervention, i.e. with FIQ score increased from at least 14% as compared to Day 00
Pain intensity | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in pain intensity measured on a Visual Analogical Scale (VAS)
Pain relief | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in pain relief measured on a VAS
Kinesiophobia index | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in kinesiophobia measured by TAMPA scale
Catastrophizing index | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in catastrophizing measured by pain catastrophizing scale (PCS)
Function impairment | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in function impairment measured by the Western Ontario and McMaster Universities Arthritis (WOMAC) scale
Fatigue | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in fatigue measured by Picot scale
Somnolence | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in somnolence measured by Epworth scale
Anxiety and depression | Week 03, Month 03, Month 06, Month 12
  Average change from baseline in anxiety and depression measured by Hospital Anxiety and Average change from baseline in anxiety and depression measured by Hospital ANxiety and Depression scale
Serious adverse reactions (SARs) | Day 00 to Month 12
  Probability of occurrence of SARs
drug consumption | Day 00, Week 03, Month 03, Month 06, Month 12
  change in drug consumption
non-drug treatment consumption | Day 00, Week 03, Month 03, Month 06, Month 12
  change in non-drug treatment consumption
Thermal outbreaks | Day 00 to Week 03
  Probability of occurrence of thermal outbreaks during the cure period
Fibromyalgia outbreaks | Week 03 to Month 12
  Probability of occurrence fibromyalgia outbreaks during remote follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DUCAMP, MD, Principal Investigator — Centre de Médecine et de Traumatologie du Sport
Locations (1):
- OTD, Dax, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diatchenko L, Nackley AG, Slade GD, Fillingim RB, Maixner W. Idiopathic pain disorders--pathways of vulnerability. Pain. 2006 Aug;123(3):226-230. doi: 10.1016/j.pain.2006.04.015. Epub 2006 Jun 13. No abstract available. PMID 16777329
- [Background] Branco JC, Saraiva F et al. Fibromyalgia Syndrom : A european epidemiological survey. Abstract Sat 0452 Eular 2005
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Haute Autorité de Santé. Le syndrome fibromyalgique de l'adulte. Rapport d'orientation. Juillet 2010. 124p
- [Background] Laroche F. Actualités de la fibromyalgie. Rev Rhum 2009;76:529-36.
- [Background] Boureau F. Modèles théoriques cognitifs et comportementaux de la douleur chronique Doul et Analg 1999 ; 4 : 265-72
- [Background] Vlaeyen JWS. Place du concept de " peur de bouger " (ré) apparition du " mal " dans l'analyse et la réhabilitation comportementale des lombalgiques chroniques. Doul et Analg, 1999 ; 4 :281-8
- [Background] Pincus T, Burton AK, Vogel S, Field AP. A systematic review of psychological factors as predictors of chronicity/disability in prospective cohorts of low back pain. Spine (Phila Pa 1976). 2002 Mar 1;27(5):E109-20. doi: 10.1097/00007632-200203010-00017. PMID 11880847
- [Background] Bannwarth B, Blotman F, Le Lay K, Boussetta S, Caubère JP, André E, Taïeb C. Prévalence of fibromyalgia : a large-scale european survey : results in France Eular 2008, Paris, THU0392
- [Background] Maugars Y, Lamotte M, De Vos C C, Girard L, Caubère JP, André E, Le Lay K, Taïeb C. Fibromyalgia : the avoied cost of the non-diagnosed patient in France. Eular 2008, Paris, THU0386
- [Background] Boureau F. in Pratique du Traitement de la Douleur. Doin ed. 1988, 402p
- [Background] Weigent DA, Bradley LA, Blalock JE, Alarcon GS. Current concepts in the pathophysiology of abnormal pain perception in fibromyalgia. Am J Med Sci. 1998 Jun;315(6):405-12. doi: 10.1097/00000441-199806000-00009. PMID 9638897
- [Background] Mountz JM, Bradley LA, Modell JG, Alexander RW, Triana-Alexander M, Aaron LA, Stewart KE, Alarcon GS, Mountz JD. Fibromyalgia in women. Abnormalities of regional cerebral blood flow in the thalamus and the caudate nucleus are associated with low pain threshold levels. Arthritis Rheum. 1995 Jul;38(7):926-38. doi: 10.1002/art.1780380708. PMID 7612042
- [Background] Valverde O, Mico JA, Maldonado R, Mellado M, Gibert-Rahola J. Participation of opioid and monoaminergic mechanisms on the antinociceptive effect induced by tricyclic antidepressants in two behavioural pain tests in mice. Prog Neuropsychopharmacol Biol Psychiatry. 1994 Oct;18(6):1073-92. doi: 10.1016/0278-5846(94)90132-5. PMID 7824761
- [Background] Van Houdenove B, Luyten P. Fibromyalgia and related syndromes characterised by stress intolerance and pain hypersensitivity: do we need a new nosology ? Curr Rheumatol Rev 2007; 3: 304-308
- [Background] Marchand S. Influences des hormones sexuelles sur les mécanismes endogens impliqués dans le développement et la persistance de la douleur. Congrès SFETD, Nantes, 2006, Douleurs, nov.2006, CS04
- [Background] Ablin JN, Cohen H, Buskila D. Mechanisms of Disease: genetics of fibromyalgia. Nat Clin Pract Rheumatol. 2006 Dec;2(12):671-8. doi: 10.1038/ncprheum0349. PMID 17133252
- [Background] Houvenagel E. Physiopathologie de la douleur de la fibromyalgie. Rev.Rhum.70(2003) :314-320
- [Background] Perrot S, Dumont D, Guillemin F, Pouchot J, Coste J; French Group for Quality of Life Research. Quality of life in women with fibromyalgia syndrome: validation of the QIF, the French version of the fibromyalgia impact questionnaire. J Rheumatol. 2003 May;30(5):1054-9. PMID 12734906
- [Background] Mothe B, Etude comparée de l'efficacité thérapeutique de l'hypnose et de la relaxation dans la fibromyalgie. Universite de Paris VIII - Vincennes - Saint-Denis. Ecole Doctorale Cognition Langage Interaction. Laboratoire de
- [Background] Gerin P, Dazord A, Cialdella P, Leizorovicz A, Boissel JP. [The questionnaire "Profile of the subjective quality of life". First data of validation]. Therapie. 1991 Mar-Apr;46(2):131-8. French. PMID 2053091
- [Background] Mailhan L. (2005). Qualité de vie après traumatisme crânien sévère. Pratiques psychologiques, 11, 343-357
- [Background] Dazord A, Mercier C, Manificat S, Nicolas J. (1995), Evaluation de la qualité de la vie : mise au point d'un instrument d'évaluation dans un contexte francophone, Revue Européenne de Psychologie Appliquée, 45, 4, 271-278
- [Background] Geenen R. Psychological approaches to management of fibromyalgia. Eular 2008, Paris, SP0124
- [Background] Mease P. Fibromyalgia syndrome: review of clinical presentation, pathogenesis, outcome measures, and treatment. J Rheumatol Suppl. 2005 Aug;75:6-21. PMID 16078356
- [Background] Coichard CG, Cabane J et al.Intérêt d'une prise en charge multidisciplinaire du patient fibromyalgique. Rev.Rhum. (2003) ; 70 :354-7
- [Background] Cedraschi C, Desmeules J, Rapiti E, Baumgartner E, Cohen P, Finckh A, Allaz AF, Vischer TL. Fibromyalgia: a randomised, controlled trial of a treatment programme based on self management. Ann Rheum Dis. 2004 Mar;63(3):290-6. doi: 10.1136/ard.2002.004945. PMID 14962965
- [Background] Goldenberg DL, Felson DT, Dinerman H. A randomized, controlled trial of amitriptyline and naproxen in the treatment of patients with fibromyalgia. Arthritis Rheum. 1986 Nov;29(11):1371-7. doi: 10.1002/art.1780291110. PMID 3535811
- [Background] Miadsi D, Juniper MD. et al. The pharmacological management of fibromyalgia syndrome in the UK primary care setting. Eular, 2008, Paris. OP0076
- [Background] Russell IJ, Kamin M, Bennett RM, Schnitzer TJ, Green JA, Katz WA. Efficacy of tramadol in treatment of pain in fibromyalgia. J Clin Rheumatol. 2000 Oct;6(5):250-7. doi: 10.1097/00124743-200010000-00004. PMID 19078481
- [Background] Biasi G, Manca S, Manganelli S, Marcolongo R. Tramadol in the fibromyalgia syndrome: a controlled clinical trial versus placebo. Int J Clin Pharmacol Res. 1998;18(1):13-9. PMID 9604730
- [Background] Bennett RM, Kamin M, Karim R, Rosenthal N. Tramadol and acetaminophen combination tablets in the treatment of fibromyalgia pain: a double-blind, randomized, placebo-controlled study. Am J Med. 2003 May;114(7):537-45. doi: 10.1016/s0002-9343(03)00116-5. PMID 12753877
- [Background] Sorensen J, Bengtsson A, Backman E, Henriksson KG, Bengtsson M. Pain analysis in patients with fibromyalgia. Effects of intravenous morphine, lidocaine, and ketamine. Scand J Rheumatol. 1995;24(6):360-5. doi: 10.3109/03009749509095181. PMID 8610220
- [Background] Trèves R, Bannwarth B, Bertin P, Javier RM, Glowinski J, Le Bars M, Perrot S. Les Recommandations de Limoges. Usage de la morphine dans les douleurs rhumatismales non cancéreuses. Douleurs, 2000, 1,1, 33-38
- [Background] Moldofsky H, Scarisbrick P. Induction of neurasthenic musculoskeletal pain syndrome by selective sleep stage deprivation. Psychosom Med. 1976 Jan-Feb;38(1):35-44. doi: 10.1097/00006842-197601000-00006. PMID 176677
- [Background] Arnold LM. Biology and therapy of fibromyalgia. New therapies in fibromyalgia. Arthritis Res Ther. 2006;8(4):212. doi: 10.1186/ar1971. PMID 16762044
- [Background] Goldenberg DL. Management of fibromyalgia syndrome. Rheum Dis Clin North Am. 1989 Aug;15(3):499-512. PMID 2672134
- [Background] Tofferi JK, Jackson JL, O'Malley PG. Treatment of fibromyalgia with cyclobenzaprine: A meta-analysis. Arthritis Rheum. 2004 Feb 15;51(1):9-13. doi: 10.1002/art.20076. PMID 14872449
- [Background] Wolfe F, Cathey MA, Hawley DJ. A double-blind placebo controlled trial of fluoxetine in fibromyalgia. Scand J Rheumatol. 1994;23(5):255-9. doi: 10.3109/03009749409103725. PMID 7973479
- [Background] Arnold LM, Hess EV, Hudson JI, Welge JA, Berno SE, Keck PE Jr. A randomized, placebo-controlled, double-blind, flexible-dose study of fluoxetine in the treatment of women with fibromyalgia. Am J Med. 2002 Feb 15;112(3):191-7. doi: 10.1016/s0002-9343(01)01089-0. PMID 11893345
- [Background] Anderberg UM, Marteinsdottir I, von Knorring L. Citalopram in patients with fibromyalgia--a randomized, double-blind, placebo-controlled study. Eur J Pain. 2000;4(1):27-35. doi: 10.1053/eujp.1999.0148. PMID 10833553
- [Background] O'Malley PG, Balden E, Tomkins G, Santoro J, Kroenke K, Jackson JL. Treatment of fibromyalgia with antidepressants: a meta-analysis. J Gen Intern Med. 2000 Sep;15(9):659-66. doi: 10.1046/j.1525-1497.2000.06279.x. PMID 11029681
- [Background] Arnold LM, Keck PE Jr, Welge JA. Antidepressant treatment of fibromyalgia. A meta-analysis and review. Psychosomatics. 2000 Mar-Apr;41(2):104-13. doi: 10.1176/appi.psy.41.2.104. PMID 10749947
- [Background] Goldenberg DL, Clauw DJ, Palmer RH, Mease P, Chen W, Gendreau RM. Durability of therapeutic response to milnacipran treatment for fibromyalgia. Results of a randomized, double-blind, monotherapy 6-month extension study. Pain Med. 2010 Feb;11(2):180-94. doi: 10.1111/j.1526-4637.2009.00755.x. Epub 2009 Dec 9. PMID 20002596
- [Background] Branco JC, Perrot S, Bragee G, Zachrisson O, Mikkelsen K, Mainguy Y, Pezous N. Milnacipran for the treatment of fibromyalgia syndrome : a European multicenter, randomized, double-blind, placebo-controlled trial. Eular 2008, Paris, THU0365
- [Background] Chappell AS, Littlejohn G, Kajdasz DK, Scheinberg M, D'Souza DN, Moldofsky H. A 1-year safety and efficacy study of duloxetine in patients with fibromyalgia. Clin J Pain. 2009 Jun;25(5):365-75. doi: 10.1097/AJP.0b013e31819be587. PMID 19454869
- [Background] Russell JI, Mease PJ, Smith TR, Kajdasz DK, Wohlreich MM, Detke MJ, Walker DJ, Chappell AS, Arnold LM. Efficacy and safety of duloxetine for treatment of fibromyalgia in patients with or without major depressive disorder: Results from a 6-month, randomized, double-blind, placebo-controlled, fixed-dose trial. Pain. 2008 Jun;136(3):432-444. doi: 10.1016/j.pain.2008.02.024. Epub 2008 Apr 18. PMID 18395345
- [Background] Zijlstra TR, Barendregt PJ, van De Laar MA. Venlafaxine in fibromyalgia: results of a randomized placebo-controlled, double-blind trial. Arthritis Rheum. 2002;46:S105
- [Background] Clère F, Henry F, Perriot M. Quelle place pour le clonazepam dans la douleur chronique ? Douleurs, vol7n°6 dec 2006 :314-317
- [Background] Arnold LM, Goldenberg DL, Stanford SB, Lalonde JK, Sandhu HS, Keck PE Jr, Welge JA, Bishop F, Stanford KE, Hess EV, Hudson JI. Gabapentin in the treatment of fibromyalgia: a randomized, double-blind, placebo-controlled, multicenter trial. Arthritis Rheum. 2007 Apr;56(4):1336-44. doi: 10.1002/art.22457. PMID 17393438
- [Background] Crofford LJ, Rowbotham MC, Mease PJ, Russell IJ, Dworkin RH, Corbin AE, Young JP Jr, LaMoreaux LK, Martin SA, Sharma U; Pregabalin 1008-105 Study Group. Pregabalin for the treatment of fibromyalgia syndrome: results of a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2005 Apr;52(4):1264-73. doi: 10.1002/art.20983. PMID 15818684
- [Background] Arnold LM, Crofford LJ, Martin SA, Young JP, Sharma U. The effect of anxiety and depression on improvements in pain in a randomized, controlled trial of pregabalin for treatment of fibromyalgia. Pain Med. 2007 Nov-Dec;8(8):633-8. doi: 10.1111/j.1526-4637.2007.00332.x. PMID 18028041
- [Background] Barrett J, Russell J, Pauer L, Whalen E, Leon T, Zeiher B. The effect of pregabalin treatment on changes in pain and sleep quality in fibromyalgia patients.Eular 2008, Paris, THU0362
- [Background] Arkfeld DG, Setoodeh KM, Abrahim J, Cole SE, Metyas S. The inability of most us patients to tolerate the recommended doses of pregabalin in the treatment of fibromyalgia ;: a case study. Elar 2008, Paris, THU0396
- [Background] Wood PB, Schweinhardt P, Jaeger E, Dagher A, Hakyemez H, Rabiner EA, Bushnell MC, Chizh BA. Fibromyalgia patients show an abnormal dopamine response to pain. Eur J Neurosci. 2007 Jun;25(12):3576-82. doi: 10.1111/j.1460-9568.2007.05623.x. PMID 17610577
- [Background] Holman AJ, Myers RR. A randomized, double-blind, placebo-controlled trial of pramipexole, a dopamine agonist, in patients with fibromyalgia receiving concomitant medications. Arthritis Rheum. 2005 Aug;52(8):2495-505. doi: 10.1002/art.21191. PMID 16052595
- [Background] Bennett RM, Clark SC, Walczyk J. A randomized, double-blind, placebo-controlled study of growth hormone in the treatment of fibromyalgia. Am J Med. 1998 Mar;104(3):227-31. doi: 10.1016/s0002-9343(97)00351-3. PMID 9552084
- [Background] Clark S, Tindall E, Bennett RM. A double blind crossover trial of prednisone versus placebo in the treatment of fibrositis. J Rheumatol. 1985 Oct;12(5):980-3. PMID 3910836
- [Background] Russell u, Bennett RM, Michalek JE. Sodium oxybrate relieves pain and improves sleep in fibromyalgia syndrome. A randomized, double-blind, placebo-controlled, multi-center clinical trial. ACR/ARHP Scientific Meeting. 2005; programm book supplement:late-breaking abstracts
- [Background] Holdcraft LC, Assefi N, Buchwald D. Complementary and alternative medicine in fibromyalgia and related syndromes. Best Pract Res Clin Rheumatol. 2003 Aug;17(4):667-83. doi: 10.1016/s1521-6942(03)00037-8. PMID 12849718
- [Background] Sarac AJ, Gur A. Complementary and alternative medical therapies in fibromyalgia. Curr Pharm Des. 2006;12(1):47-57. PMID 16454724
- [Background] Perrot S, Maheu E, Javier RM, Eschalier A, Coutaux A, LeBars M, Bertin P, Bannwarth B, Treves R. Guidelines for the use of antidepressants in painful rheumatic conditions. Eur J Pain. 2006 Apr;10(3):185-92. doi: 10.1016/j.ejpain.2005.03.004. Epub 2005 Apr 18. PMID 16490727
- [Background] Journal Officiel de la République Française, 9 août 2006. Arrêté du 1er août 2006 portant approbation d'un avenant à la convention nationale thermale.
- [Background] Thermalisme et santé publique vers de nouvelles convergences. Livre Blanc CNETH 2008.
- [Background] Rapport 2011 du Conseil National du Tourisme pour le Ministre chargé du Tourisme " réflexions et propositions sur la diversification des stationsThermales ".
- [Background] Bellometti S, Galzigna L. Function of the hypothalamic adrenal axis in patients with fibromyalgia syndrome undergoing mud-pack treatment. Int J Clin Pharmacol Res. 1999;19(1):27-33. PMID 10450540
- [Background] Adler GK, Geenen R. Hypothalamic-pituitary-adrenal and autonomic nervous system functioning in fibromyalgia. Rheum Dis Clin North Am. 2005 Feb;31(1):187-202, xi. doi: 10.1016/j.rdc.2004.10.002. PMID 15639063
- [Background] McLean SA, Williams DA, Harris RE, Kop WJ, Groner KH, Ambrose K, Lyden AK, Gracely RH, Crofford LJ, Geisser ME, Sen A, Biswas P, Clauw DJ. Momentary relationship between cortisol secretion and symptoms in patients with fibromyalgia. Arthritis Rheum. 2005 Nov;52(11):3660-9. doi: 10.1002/art.21372. PMID 16258904
- [Background] Donmez A, Karagulle MZ, Tercan N, Dinler M, Issever H, Karagulle M, Turan M. SPA therapy in fibromyalgia: a randomised controlled clinic study. Rheumatol Int. 2005 Dec;26(2):168-72. doi: 10.1007/s00296-005-0623-9. Epub 2005 Jun 17. PMID 15965635
- [Background] Zijlstra TR, van de Laar MA, Bernelot Moens HJ, Taal E, Zakraoui L, Rasker JJ. Spa treatment for primary fibromyalgia syndrome: a combination of thalassotherapy, exercise and patient education improves symptoms and quality of life. Rheumatology (Oxford). 2005 Apr;44(4):539-46. doi: 10.1093/rheumatology/keh537. Epub 2005 Feb 3. PMID 15695301
- [Background] Fioravanti A, Perpignano G, Tirri G, Cardinale G, Gianniti C, Lanza CE, Loi A, Tirri E, Sfriso P, Cozzi F. Effects of mud-bath treatment on fibromyalgia patients: a randomized clinical trial. Rheumatol Int. 2007 Oct;27(12):1157-61. doi: 10.1007/s00296-007-0358-x. Epub 2007 May 23. PMID 17520260
- [Background] C. Robert, Fibromyalgie et cures thermales. Journée d'Automne de l'Institut du thermalisme Dax 27/11/2009
- [Background] Carville SF, Arendt-Nielsen L, Bliddal H, Blotman F, Branco JC, Buskila D, Da Silva JA, Danneskiold-Samsoe B, Dincer F, Henriksson C, Henriksson KG, Kosek E, Longley K, McCarthy GM, Perrot S, Puszczewicz M, Sarzi-Puttini P, Silman A, Spath M, Choy EH; EULAR. EULAR evidence-based recommendations for the management of fibromyalgia syndrome. Ann Rheum Dis. 2008 Apr;67(4):536-41. doi: 10.1136/ard.2007.071522. Epub 2007 Jul 20. PMID 17644548
- [Background] Simon D, Traynard PY, Bourdillon F, Gagnaire R, Grimaldi A. Education thérapeutique, prévention et maladies chroniques. Masson. 2ème édition 2011.
- [Background] Résultats de l'étude TNS Healthcare auprès de 112 000 curistes 2006 source CNETH 1 rue Cels 75016 Paris.
- [Background] Ducamp Ph.Le thermalisme peut-il être le lieu idéal de la prise en charge des patients fibromyalgiques ? Mémoire de fin d'études du diplôme universitaire d'éducation thérapeutique de formation et de coordination d'équipe. UMFMC Université Bordeaux Segalen 2012.
- [Background] Ducamp Ph. Journées Nationales du thermalisme Luchon Nov 2012. La place des médecins thermaux dans l'éducation thérapeutique.
- [Background] Haute Autorité de Santé. Guide méthodologique
- [Background] Sichère P. Fibromyalgie, éducation thérapeutique, thermalisme. Mémoire de fin d'études et de formation à l'éducation thérapeutique IPCEM. IPCEM 2012.
- [Background] Sichère P, Ducamp P. Fibromyalgie, éducation thérapeutique, thermalisme. Congrès national de la Société Française de Rhumatologie (M149) Paris 8-12 décembre 2012.
- [Background] Ducamp Ph. Fibromyalgie, éducation thérapeutique et thermalisme. La presse thermale et climatique, Nov 2011.
- [Background] Sichère P. Evaluation, diagnostics, traitements. Douleurs 2012; 13: 244-6: Douleurs et thermalisme: questions posées au Dr Philippe Ducamp.
- [Background] Sichère P et Ducamp P. Éducation thérapeutique, fibromyalgie et thermalisme. Douleurs 2013; 14: 22-9.
- [Background] Françon A, Queneau P. Quelle place pour la crénothérapie dans la fibromyalgie ? Abrégé " Médecine thermale. Faits et preuves ". P. Queneau et coll. Edition Masson 2000, p 75-77
- [Background] Françon A. Fibromyalgie et thermalisme. N°125-14-janvier 2010-reflexions Rhumato.p15-18
- [Background] D'Ivernois JF, Gagnayre R. Propositions pour l'évaluation de l'éducation thérapeutique. In ADSP, n°58, mars 2007
- [Background] Foucaud J, Bury JA, Balcou-Debussche M, Eymard C. Education thérapeutique du patient : Modèles, pratiques et évaluation. Dir. Saint Denis INPES, collection Santé en Action, 2010 : 412p.
- [Background] Roberts PJ, Torgerson DJ, BMJ 2002
- [Background] Perrot S, Bouhassira D, Fermanian J; CEDR (Cercle d'Etude de la Douleur en Rhumatologie). Development and validation of the Fibromyalgia Rapid Screening Tool (FiRST). Pain. 2010 Aug;150(2):250-256. doi: 10.1016/j.pain.2010.03.034. Epub 2010 May 21. PMID 20488620
- [Background] Huet AG. Une expérience d'Art-Thérapie, à dominante danse, auprès des personnes fibromyalgiques. Université François Rabelais ; UFR médecine Tours. 2011.
- [Background] Graber-Duvernay B. Dix ans de surveillance épidémiologique des pneumopathies à Aix-les-Bains (1990 - 1999). Presse Therm Clim 2001; 138: 13-25
- [Background] Gerbaud L, Maire A, Devaux I, Chadès C, Riguidel Ph, Vidal A, Glanddier Ph Y. La surveillance des incidents infectieux chez les curistes thermaux en auvergne synthèse de 8 années d'expérience de réseaux sentinelles. Presse Therm Clim 2001; 138: 41-50
- [Background] Fournet D. La surveillance des incidents infectieux chez les curistes de Balaruc-les-Bains. Presse Therm Clim 2001; 138: 51-53
- [Background] Françon A, Graber-Duvernay B, Forestier R, Palmer M. Incidence des évènements infectieux dans une population de curistes présumés vulnérables. Presse Therm Clim 2001; 138: 55-65
- [Background] Leclerc H. Bactériologie de Pseudomonas aeruginosa. Presse Therm Clim 2002; 139: 9-13
- [Background] Ruimy R. Pathogénicité de Pseudomonas aeruginosa en dehors de la mucoviscidose. Presse Therm Clim 2002; 139: 15-21
- [Background] Tancréde-Bohin E. Pseudomonas et infections cutanées. Presse Therm Clim 2002; 139: 23-28
- [Background] Barry B. Pseudomonas aeruginosa et infections ORL. Presse Therm Clim 2002; 139: 29-33
- [Background] Graber-Duvernay B. Pseudomonas aeruginosa et infections broncho-pulmonaires. Presse Therm Clim 2002; 139: 35-40
- [Background] Morin J.P, Graber-Duvernay B. Surveillance des pseudomonas et expériences de désinfection. Presse Therm Clim 2002; 139: 41-51
- [Background] Hartemann Ph. Quelles mesures préconiser pour une gestion raisonnée du risque dû a Pseudomonas aeruginosa ? Presse therm climat 2002; 139: 53-57
- [Background] Nguyen Ba B, Dubourg K, Pécastaings S, Optimisation de la lutte contre les légionnelles et autres opportunistes dans les réseaux d'eau minérale naturelle, grâce à un pilote "eau thermale". Press Therm Clim 2006;143:7-123
- [Background] R Forestier, A Françon, Graber-Duvernay B, Palmer M, sevez JF, Guillemot A, BErnard JP, Souchon JF, Gerrud S, Le Provost C, Joly J, Rogeaux O, Deschamps O. Incidence des événements infectieux survenus en cure thermale dans une population de curistes présu- més vulnérables : étude contrôlée longitudinale sur 738 patients. Press Therm Clim 2008;145:9-21
- [Background] Dubourg K, Grégoire P, Lagière J. La désinfection des piscines thermales de Dax. Press Therm Clim 2008;145:61-71
- [Background] Ducamp P. Fibromyalgie et thermalisme. 10ème Congrès National de la Fibromyalgie FNAFF. Nîmes, 13 octobre 2012.
- [Background] Grille OPTIMON évaluant le risque patient dans les études de recherche clinique institutionnelles
- [Background] Sous-groupe de travail Qualité de la promotion - Plan de monitoring adapté - DRCI Hospices Civils de Lyon. Elaboration du plan de monitoring adapté pour une recherche biomédicale à promotion institutionnelle
- [Background] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473